CLINICAL TRIAL: NCT01827020
Title: Effect of Ketamine Addition to Lidocaine for Postoperative Pain Management in Rhinoplasty
Brief Title: Effect of Ketamine Addition to Lidocaine in Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mukadder Sanli, MD, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mukadder
Record Dates: First submitted 2013-03-28; First posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Nose Deformities, Acquired
MeSH Terms: conditions — Nose Deformities, Acquired | interventions — Ketamine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group L (number of participants=30) (Active Comparator): After standard anesthesia induction and before surgery, patients will receive submucosal infiltration of 12 mL lidocaine 2%, 1mg/kg into nasal cavity.
  Interventions: Drug: Lidocaine 2 %
- Group K (number of participants=30) (Active Comparator): After standard anesthesia induction and before surgery, patients will receive submucosal infiltration of 12 mL ketamine 0.5 mg/kg plus lidocaine 2% 1 mg/kg of the intranasal cavity.
  Interventions: Drug: Ketamine plus Lidocaine
- Group S (number of participants=30) (Placebo Comparator): After standard anesthesia induction and before surgery, patients will receive submucosal infiltration of saline 12 mL into intranasal cavity.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine 2 % — 12 mL lidocaine 2% 1mg/kg
  Other Names: preincisional infiltration of lidocaine
  Arms: Group L (number of participants=30)
Drug: Ketamine plus Lidocaine — ketamine 0.5 mg/kg + Lidocaine 2% 1 mg/kg in total volume of 12 mL
  Other Names: preincisional infiltration of ketamine plus lidocaine
  Arms: Group K (number of participants=30)
Drug: Saline — 12 mL saline (0.9% isotonic solution)
  Other Names: preincisional infiltration of saline
  Arms: Group S (number of participants=30)

SUMMARY:
The purpose of this study is to determine whether subanesthetic ketamine addition to lidocaine decreases postoperative pain scores in infiltration anesthesia during rhinoplasty.

DETAILED DESCRIPTION:
In rhinoplasty operations local infiltration anesthesia uses for surgery insight and patient comfort. The investigators designed this study to prolonged the time of infiltration block and preventive analgesia. So, before operation, study drugs will infiltrate to the submucosa of intranasal cavity. Then, surgeon and patient satisfaction, postoperative analgesic demand, postoperative pain scores and side effects will determine.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective rhinoplasty operation under general anesthesia
* Patients with ASA (American Society of Anesthesiology) class I
* Patients between 18-50 years old

Exclusion Criteria:

* Age <18 and >50
* ASA > II
* Preexisting neurological or psychiatric illness
* Systemic diseases (diabetes mellitus, hypertension, coronary heart disease...)
* Having a history of chronic pain and receiving chronic analgesia therapy
* Having a history of drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores on the Visual Analogue Scale | 24 hours
  Pain scores will examine with Visual analogue scale (VAS, 0-100) in the first 24 hours of postoperative period. The examination will repeated in different time period(5.min, 15.min, 30.min, 1 h, 2h,4.h, 6.h, 8.h, 16.h, 24.h). Patients that have VAS>40 will receive 1mg/kg tramadol.

SECONDARY OUTCOMES:
Patient satisfaction | 24 hour
  At the end of postoperative 24 h, the patient satisfaction will examine by a score as (1 poor, 2 middle, 3 good, 4 perfect)
Analgesic demand | 24 hour
  At the first day of postoperative period, analgesic requirement will record. When Visual analogue scale > 40, intravenous 1 mg/kg tramadol bolus will give.

OTHER OUTCOMES:
Number of participants with adverse effects as a measure of safety and tolerability | 24 hour
  Sedation, nausea and vomiting, dizziness, and hallucination will examine as an adverse effect in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mukadder Sanli, MD, Principal Investigator — Turgut Ozal Medical Center
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Honarmand A, Safavi M, Karaky H. Preincisional administration of intravenous or subcutaneous infiltration of low-dose ketamine suppresses postoperative pain after appendectomy. J Pain Res. 2012;5:1-6. doi: 10.2147/JPR.S26476. Epub 2011 Dec 30. PMID 22328829